CLINICAL TRIAL: NCT01707043
Title: Patient Preference of Taclonex Ointment to Taclonex Scalp Suspension in Adult Subjects With Psoriasis Vulgaris
Acronym: PSTaclonex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB00021361
Record Dates: First submitted 2012-10-09; First posted 2012-10-15 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Plaque Psoriasis
Keywords: plaque psoriasis; taclonex; crossover
MeSH Terms: interventions — betamethasone dipropionate, calcipotriol drug combination; calcipotriene; Suspensions

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Taclonex Ointment First (Active Comparator): All subjects will use Taclonex® (calcipotriene 0.005% and betamethasone dipropionate 0.064%) Ointment once daily for three days to affected areas, then switch to Taclonex Scalp® (calcipotriene 0.005% and betamethasone dipropionate 0.064%) Topical Suspension once daily to affected areas for three days
  Interventions: Drug: Taclonex
- Taclonex Scalp Suspension first (Active Comparator): All subjects will use Taclonex Scalp® (calcipotriene 0.005% and betamethasone dipropionate 0.064%) Topical Suspension once daily to affected areas for three days, then switch to Taclonex® (calcipotriene 0.005% and betamethasone dipropionate 0.064%) Ointment once daily for three days to affected areas,
  Interventions: Drug: Taclonex

INTERVENTIONS:
Drug: Taclonex — Subjects will be evaluated at baseline, Day 3 and Day 6 (or end of study).
  Other Names: Taclonex® Ointment; (calcipotriene 0.005% betamethasone dipropionate 0.064%); Taclonex Scalp®; (calcipotriene 0.005% and betamethasone dipropionate 0.064%); Topical Suspension

SUMMARY:
This is an open label, investigator-blinded, cross over, prospective, single center study of subjects with plaque psoriasis. Taclonex® (calcipotriene 0.005% and betamethasone dipropionate 0.064%) Ointment and Taclonex Scalp® (calcipotriene 0.005% and betamethasone dipropionate 0.064%) Topical Suspension will each be applied topically once daily.

The primary objective is to assess the patient preference for Taclonex® (calcipotriene 0.005% and betamethasone dipropionate 0.064%) Ointment compared to Taclonex Scalp® (calcipotriene 0.005% and betamethasone dipropionate 0.064%) Topical Suspension in the treatment of plaque psoriasis.

DETAILED DESCRIPTION:
* Following satisfaction of entry criteria, all subjects at the Baseline/Screening visit will be randomized 1:1 to receive either Taclonex® (calcipotriene 0.005% and betamethasone dipropionate 0.064%) Ointment or Taclonex Scalp® (calcipotriene 0.005% and betamethasone dipropionate 0.064%) Topical Suspension to use once daily for three days to affected areas of the body, excluding face and intertriginous areas. Subjects will be aware of which product they are using. Investigators will remain blinded.
* Subjects will be randomized to use either the ointment or the scalp suspension for the first three day treatment period, then cross over to use the other product for second three day treatment period.
* Each medication will be used within its FDA-approved label for the treatment of plaque psoriasis in subjects aged 18 and older. Subjects may not treat areas of the face, axilla or groin in this study.
* At the Day 3 and Day 6 visits the subjects will complete a questionnaire about their psoriasis treatment preferences.
* Pregnancy tests will be done on females of childbearing potential at Baseline/Screening.
* Adverse events will be monitored at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, age 18 or older, in good health.
* Subject has plaque-type psoriasis- no history of or current pustular, erythrodermic or guttate psoriasis.
* Subject is capable of understanding and willing to provide a signed and dated written voluntary informed consent before any protocol specific procedures are performed.
* The percentage of overall body surface involvement is between 1-10% on the trunk or extremities and is amenable to topical treatment with less than 100g of topical medication per week.
* The subject has an investigator global assessment of mild to moderate plaque psoriasis (severity index between 2 and 3 on a 5 point scale).
* The subject is able to complete the study and comply with study instructions, including attending all study visits.
* If a female subject of childbearing potential, subject has a negative urine pregnancy test. Sexually active women of childbearing potential participating in the study must have been using a medically acceptable form of contraception (which includes barrier methods, oral contraception, injectable or implantable methods, or intrauterine devices) for at least three months prior to entry into the study. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant. Abstinence is considered an acceptable method of contraception.

Exclusion Criteria:

* Subject has used experimental drugs or devices at least one month prior to Baseline.
* Subject has used systemic corticosteroid, phototherapy, retinoids, methotrexate, cyclosporine, or other immunosuppressive agents or biologics therapy (ie, alefacept, etanercept, efalizumab) within four weeks of Baseline.
* Subject has used topical therapy, corticosteroid therapy, topical vitamin D analog or calcineurin inhibitors or , tazarotene within two weeks prior to the Baseline visit (eg, tar, anthralin, salicylic acid, lactic acid, urea preparations).
* Subject has other serious skin disorder or any chronic medical condition that is not well controlled.
* Subject has clinically relevant abnormal vital signs or findings on the physical examination.
* Subject has major illness within 30 days prior to the Baseline visit.
* Subject has history of any immunocompromising disease.
* Subject is pregnant or nursing. Pregnant and nursing females will not be allowed in the study, and females of childbearing potential will have a pregnancy test at Baseline.
* Subject has a skin condition or disease that may require concurrent therapy or may confound the evaluation; a history of hypersensitivity to any of the formulation components; or atopic dermatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve R Feldman, M.D, Ph.D., Principal Investigator — Wake Forest University Health Sciences; Alan B Fleischer, Jr, M.D., Principal Investigator — Wake Forest University Health Sciences; Adele R Clark, PA-C, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Taclonex Scalp Suspension First, Then Taclonex Ointment: All subjects will use Taclonex Scalp® (calcipotriene 0.005% and betamethasone dipropionate 0.064%) Topical Suspension once daily to affected areas of psoriasis for three days.
  Subjects will then cross over to use Taclonex ointment for 3 days. There is no washout between products.
- Taclonex Ointment First, Then Taclonex Scalp Suspension: All subjects will use Taclonex Ointment to psoriasis twice daily for 3 days Subjects will then cross over to use Taclonex Scalp Suspension for 3 days.There is no washout between products.
Period: Overall Study
Arm/Group | Taclonex Scalp Suspension First, Then Taclonex Ointment | Taclonex Ointment First, Then Taclonex Scalp Suspension
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Taclonex Scalp Suspension First, the Taclonex Ointment: All subjects will use Taclonex Scalp Suspension first to psoriasis twice daily for 3 days Subjects will then cross over to use Taclonex Ointment for 3 days.There is no washout between products.
- Taclonex Ointment First Then Taclonex Scalp Suspension: All subjects will use Taclonex Ointment to psoriasis twice daily for 3 days Subjects will then cross over to use Taclonex Scalp Suspension for 3 days.There is no washout between products.
- Total: Total of all reporting groups
Arm/Group | Taclonex Scalp Suspension First, the Taclonex Ointment | Taclonex Ointment First Then Taclonex Scalp Suspension | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Full Range); unit: years] | 49.5 [29 to 64] | 47 [33 to 63] | 48 [29 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 8 | 18
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Subjective Subject Preference Survey for the First Treatment Session
Description: Subjective Subject Preference Survey The Subjective Subject Preference Survey consist of 15 questions relating to patients preference of study drug. The survey includes questions such as how the medication feels to touch, how greasy it is, and time it takes to apply. The final question asks patients to rate the overall appeal of the vehicle. Questions are scored on a 7-point scale, where a score of 1 is extremely unpleasant, 4 is neutral, and a score of 7 is extremely appealing. Total preference score based on the Subjective Subject Preference Survey could range from 15-105.
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Taclonex Scalp Suspension First Then Taclonex Ointment: All subjects will use Taclonex Scalp® (calcipotriene 0.005% and betamethasone dipropionate 0.064%) Topical Suspension once daily to affected areas of psoriasis for three days.
  Subjects will then cross over to use Taclonex ointment for 3 days. There is no washout between products.
- Taclonex Ointment First, Then Taclonex Scalp Suspension: All subjects will use Taclonex Scalp® (calcipotriene 0.005% and betamethasone dipropionate 0.064%) Ointment once daily to affected areas of psoriasis for three days.
  Subjects will then cross over to use Taclonex Suspension for 3 days. There is no washout between products.
Arm/Group | Taclonex Scalp Suspension First Then Taclonex Ointment | Taclonex Ointment First, Then Taclonex Scalp Suspension
Number analyzed (Participants) | 10 | 10
units on a scale | 81.1 (18.4) | 77.6 (21.2)

2. Primary Outcome: Subjective Subject Preference Survey for the Second Treatment Session
Description: as for outcome 1
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taclonex Scalp Suspension First Then Taclonex Ointment | Taclonex Ointment First, Then Taclonex Scalp Suspension
Number analyzed (Participants) | 10 | 10
units on a scale | 78.9 (22.8) | 69.4 (17.6)

ADVERSE EVENTS:
Time Frame: data collected at each visit over one week
Groups:
- Taclonex Ointment: All subjects will use Taclonex® (calcipotriene 0.005% and betamethasone dipropionate 0.064%) Ointment once daily for three days to affected areas In this arm, subject will give a preference rating for Taclonex Ointment
- Taclonex Scalp Suspension: All subjects will use Taclonex Scalp® (calcipotriene 0.005% and betamethasone dipropionate 0.064%) Topical Suspension once daily to affected areas for three days.
  In this arm, subjects will give a preference rating for the Suspension
Arm/Group | Taclonex Ointment | Taclonex Scalp Suspension
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days